CLINICAL TRIAL: NCT00116454
Title: A Randomized and Multicenter Trial for Hepatocellular Carcinoma Adjuvant Treatment by Lipiocis
Brief Title: Trial for Hepatocellular Carcinoma Adjuvant Treatment by Lipiocis
Acronym: Lipiocis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004-003883-31; ANRS HC06 LIPIOCIS (Other: ANRS)
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Carcinoma, Hepatocellular; Hepatitis, Viral, Human
Keywords: Carcinoma, Hepatocellular; Viral Hepatitis, Alcoholic Hepatitis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis, Viral, Human; Hepatitis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lipiocis group (Experimental): intra-arterial hepatic administration, one 2200 MBQ dose, duration of treatment 1 week
  Interventions: Drug: 131 I-lipiodol
- control group (No Intervention): group untreated

INTERVENTIONS:
Drug: 131 I-lipiodol — intra-arterial hepatic administration of Lipiocis will occur, 11 to 12 weeks after the initial curative treatment
  Other Names: Lipiocis
  Arms: lipiocis group

SUMMARY:
The recurrence of hepatocellular carcinoma (HCC), two years after curative treatment is high, about 40% - 50%. Recently, it has been shown that intra-arterial radioactive lipiodol (Lipiocis®) could reduce the recurrence of cancer and increase the survival after resection of HCC developed on cirrhosis B. The aim of the present trial is to investigate the effect of Lipiocis® in preventing recurrence after curative treatment of HCC in patients with viral or alcoholic hepatitis related cirrhosis by surgical or percutaneous ablation.

DETAILED DESCRIPTION:
The usual therapeutic approaches of early hepatocellular carcinoma (HCC) are partial hepatectomy or percutaneous ethanol injection. However, these therapeutic procedures do not suppress the cirrhotic liver tissue which represents a major risk factor for recurrence and/or occurrence of a second tumor in the liver. Recently, it has been shown that intra-arterial radioactive lipiodol (Lipiocis®) could reduce the recurrence of cancer and increase the survival after resection of HCC developed on cirrhosis B. The aim of the present randomized and multicenter trial is to investigate the effect of iodine-131-labelled lipiodol (131I-lipiodol = Lipiocis®) in preventing recurrence after curative treatment of HCC (hepatocellular carcinoma) in patients with viral or alcoholic hepatitis related cirrhosis by surgical or percutaneous ablation. The period of this study will be 3 years including 1 year for the enrollment and 2 years for the follow-up. Fifty patients will receive one 2200 MBq dose of Lipiocis and 50 patients will not be treated by Lipiocis (control group). The intra-arterial hepatic administration of Lipiocis will occur 11 to 12 weeks after the initial curative treatment.

The inclusion criteria are as follows : 1) men or women, aged between 18 and 75 years old, with cirrhosis or chronic hepatitis associated with C, B, delta infection or alcool intake or both and confirmed by liver biopsy and 2) one or two HCC nodules treated by surgical or percutaneous ablation (ethanol, acetic acid 50% or radiofrequency).

The efficacy of the initial curative treatment will be assessed by the following criteria: alpha-fetoprotein concentration below 25ng/ml, no progression in size of the tumour demonstrated by ultrasonography and no arterial hypervascularization on CT scan imaging.

The patients with the following criteria will be excluded: co-infection with HIV (Human Immunodeficiency Virus)associated with a CD count <200/mm3 and a viral charge >5000 HIV RNA copies/ml, documented iodine intolerance, respiratory disease, decompensated cirrhosis (Child-Pugh score over or equal 8), bilirubin concentration over 51µmol/l, portal or hepatic vein thrombosis, extra-hepatic metastasis, excessive alcohol intake (over 50g per day), blood platelet count below 50,000/mm3, neutrophil count below 1500/mm3, creatininemia over 120µmol/l, other severe concurrent disease, previous treatment for hepatocellular carcinoma and women who can be pregnant or breastfeeding.

The main endpoint will be to determine whether the Lipiocis® treatment reduces the percentage of recurrence from 50% to 20% at 24 months. The secondary end-points will be the overall survival, the survival without recurrence of the primary tumor, the survival without new tumor, the deterioration of hepatocellular function and the side effects of the Lipiocis® treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women , aged between 18 and 75 years old
* Cirrhosis or chronic hepatitis associated with C, B, delta infection or alcool intake or both and confirmed by liver biopsy
* One or two HCC nodules treated by surgical or percutaneous ablation (ethanol, acetic acid 50% or radiofrequency).
* The efficacy of the initial curative treatment will be assessed by the following criteria: alpha-fetoprotein concentration < or equal 25ng/ml, no progression in size of the tumour demonstrated by ultrasonography and no arterial hypervascularization on CT scan imaging

Exclusion Criteria:

* HIV coinfection associated with a CD count<200/mm3 and a viral charge>5000 HIV RNA copies/ml
* Documented iodine intolerance
* Respiratory insufficiency
* Decompensated cirrhosis (Child-Pugh score over 8)
* Bilirubin concentration over 51 µmol/l
* Portal or hepatic vein thrombosis
* Extra-hepatic metastasis
* Excessive alcohol intake (over 50g per day)
* Blood platelet count below 50000/mm3
* Neutrophil count above 1500/mm3
* Creatininemia over 120µmol/l
* Myocardial infarction or rhythm disorders
* Psychiatric disease with hospitalization
* Previous treatment for hepatocellular carcinoma
* Pregnant or breastfeeding
* Treatment with interferon and/or ribavirin 3 months before inclusion
* Treatment with tamoxifen or somatostatin analogs or systemic chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
to determine if the Lipiocis treatment decreases the % of tumoral recurrence after 24 months, judged on the rise of alpha-fetoprotein and the reappearance of one or more tumours on the hepatic CT scan | at 24 Months

SECONDARY OUTCOMES:
overall survival | at 24 months
recurrence-free survival | at 24 months
treatment toxicity | at 24 months
Deterioration of the hepatocellular function | at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rosmorduc, MD, Principal Investigator — Hopital Saint Antoine SERVICE D'HEPATOLOGIE; Fabrice Carrat, MD, Study Director — INSERM U 444 FACULTE DE MEDECINE ST ANTOINE
Locations (1):
- Service d'Hépatologie Hôpital Saint Antoine, Paris, France

REFERENCES:
- See also: Related Info — http://www.anrs.fr